CLINICAL TRIAL: NCT01122667
Title: A Single-Dose Study to Investigate the Pharmacokinetics of MK0859 in Subjects With Impaired Renal Function
Brief Title: Pharmacokinetics of Anacetrapib (MK0859) in Subjects With Impaired Renal Function (MK-0859-038)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0859-038; MK0859-038
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Dyslipidemia
Keywords: Renal Insufficiency
MeSH Terms: conditions — Dyslipidemias; Renal Insufficiency | interventions — anacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1 - Panel A (Experimental): Subjects with severe renal impairment
  Interventions: Drug: anacetrapib
- Part 1 - Panel B (Experimental): Healthy matched control subjects
  Interventions: Drug: anacetrapib
- Part 2 - Panel C (Experimental): Subjects with moderate renal impairment
  Interventions: Drug: anacetrapib
- Part 2 - Panel D (Experimental): Healthy matched control subjects
  Interventions: Drug: anacetrapib
- Part 2 - Panel E (Experimental): Subjects with mild renal impairment
  Interventions: Drug: anacetrapib
- Part 2 - Panel F (Experimental): Healthy matched control subjects
  Interventions: Drug: anacetrapib

INTERVENTIONS:
Drug: anacetrapib — single dose administration of anacetrapib (MK0859) 100 mg oral tablet

SUMMARY:
This study will evaluate the Area Under the Curve (AUC(0 to infinity)) of anacetrapib in subjects with impaired renal function and healthy matched control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of reproductive potential test negative for pregnancy and agree to use two acceptable methods of birth control throughout the study
* Subject is in good health
* If Subject is a smoker, smoking is limited to no more than 10 cigarettes per day

Exclusion Criteria:

* Subject has a history of stroke, chronic seizures or major neurological disorder
* Subject has a history of cancer
* Subject is unable to refrain from or anticipates the use of any prescription or non-prescription medication during the study
* Subject consumes excessive amounts of alcohol or caffeine
* Subject has had major surgery, donated blood or participated in another investigational study within the past 4 weeks
* Subject is a nursing mother
* Subject has had a kidney removed or has a functioning renal transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC(0 to infinity)) of anacetrapib | through 168 hours post dose

SECONDARY OUTCOMES:
Safety and tolerability of a single dose administration of 100mg anacetrapib, measured by the number of clinical and laboratory adverse events | through 14 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lauring B, Li XS, Liu Y, Corr C, Lazarus N, Cote J, Larson P, Levonas AO, Lasseter KC, Preston RA, Smith WB, Lai E, Wagner JA. Influence of renal and hepatic impairment on the pharmacokinetics of anacetrapib. J Clin Pharmacol. 2014 Nov;54(11):1247-55. doi: 10.1002/jcph.320. Epub 2014 Jun 6. PMID 24782116